CLINICAL TRIAL: NCT00596414
Title: Sedation and Analgesia for Transjugular Liver Biopsy: A Randomized Double Blind Placebo Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Olivier Le Moine, MD, PhD, Erasme University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BHTJ-1; BHTJ-1
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-12

CONDITIONS: Cirrhosis; Chronic Hepatitis; Anxiety
Keywords: liver; biopsy
MeSH Terms: conditions — Fibrosis; Hepatitis, Chronic; Anxiety Disorders | interventions — Midazolam; Meperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Procedure: transjugular liver biopsy; Drug: placebo
- 2 (Experimental): midazolam
  Interventions: Procedure: transjugular liver biopsy; Drug: midazolam
- 3 (Experimental): midazolam + pethidine
  Interventions: Procedure: transjugular liver biopsy; Drug: midazolam + pethidine

INTERVENTIONS:
Procedure: transjugular liver biopsy — liver biopsy through the transjugular route with hepatic-venous pressure gradient measurement
Drug: placebo
  Arms: 1
Drug: midazolam
  Arms: 2
Drug: midazolam + pethidine
  Arms: 3

SUMMARY:
Transjugular liver catheterisation allows the measurement of hepatic venous pressure gradient (HVPG) and the sampling of liver tissue but patient's tolerance to the procedure is unknown. The aim of this study was to assess tolerance to transjugular hepatic liver biopsy with or without conscious sedation/analgesia.

DETAILED DESCRIPTION:
Consecutive patients undergoing transjugular liver biopsy will be randomly assigned to receive either placebo or midazolam (0.02 mg/kg) or 0.02 mg/kg midazolam combined with 1 mg/kg pethidine before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* suspected liver disease
* known liver disease

Exclusion Criteria:

* liver transplants
* hepatocellular carcinoma
* hypersensitivity or allergy to benzodiazepines or morphinic derivatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2003-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Patient tolerance to the procedure | 1 hour after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme - Dpt of Gastroenterology, Brussels, Belgium